CLINICAL TRIAL: NCT07177690
Title: A Study of the Impact of Penicillin Allergy on Antimicrobial Resistance and ouTcomes
Acronym: IMPAART
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Jonathan Sandoe, Associate Clinical Professor, University of Leeds
Other Study IDs: Version 1. 3 25/01/2022
Record Dates: First submitted 2025-07-22; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Penicillin Allergy; Antimicrobial Drug Resistance; AMR
Keywords: penicillin allergy; AMR; Antimicrobial resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Workstream 1: PEACH Study participants: Adults and adolescents 16 years old and older, admitted to hospital between 1/2/20 and 30/06/20 with a positive SARS-CoV-2 test.
- Workstream 2 exposure group: Adult patients with a penicillin allergy attending immunology clinics at Leeds Teaching Hospitals, UK
- Workstream 2 comparator group: Adult patients without a penicillin allergy attending immunology clinics at Leeds Teaching Hospitals, UK
- Workstream 3 exposure group: Participants enrolled in the ALABAMA trial who underwent penicillin allergy testing
- Workstream 3 comparator group: Participants enrolled in the ALABAMA trial who had usual care only (i.e. did not undergo penicillin allergy testing)

SUMMARY:
Penicillin allergy is one of the commonest reported allergies. The presence of a penicillin allergy record in a patients notes leads to the avoidance of recommended first-line penicillin antibiotics and the use of alternative non-penicillin antibiotics which can be less effective, have more side effects and have a greater propensity to drive antimicrobial resistance (AMR). Most patients with penicillin allergy records do not have a true allergy when they are tested by a specialist, so many patients are denied the best antibiotics because of an incorrect penicillin allergy record.

The study will investigate how having a penicillin allergy impacts on treatment for patients who need antibiotics when they are hospitalised with COVID-19 and how penicillin allergy affects AMR.

Antibiotic use is the main driver of AMR, antibiotic use can also disrupt the bacteria that normally live in our guts and mouths. These bacterial communities also known as the gastrointestinal (GI) and oral microbiome respectively, help us digest food and prevent infections. Antibiotic use can 'kill off' these harmless bacteria and lead to an increase in bacteria which have genes that make them resistant to antibiotics (antibiotic resistance genes). The study investigators believe that patients with penicillin allergy are likely to have a greater number of antibiotic resistance genes in their oral and GI microbiomes, ans that this will make it more likely that they will fail antibiotic treatment and will increase their risk of transmitting resistance to others.

The study objectives are:

1. To determine how penicillin allergy impacts on clinical outcomes in patients admitted with COVID-19
2. To find out if AMR genes in the oral microbiome of people with a penicillin allergy record are different to those without a penicillin allergy record
3. To investigate whether AMR genes are lost in patients who have an incorrect penicillin allergy label removed

DETAILED DESCRIPTION:
Study hypothesis:

Patients with a penicillin allergy record are more likely to have resistance to non-penicillin antibiotics in their normal flora and that this will increase their risk of treatment failure with non-penicillin antibiotics. In particular, penicillin allergic patients admitted with COVID-19 who have bacterial infections will have an increased risk of treatment failure and poor outcomes.

Study design:

This research will be conducted in three separate but complementary workstreams:

Workstream 1 will include secondary analysis of data collected as a part of the Procalcitonin Evaluation of Antibiotic use in COVID-19 Hospitalised patients (PEACH) study (ISRCTN66682918) to determine how penicillin allergy impacts on antibiotic use and clinical outcomes in patients admitted with COVID-19. The PEACH study was a multi-centre, retrospective, observational, cohort study using patient-level clinical data which investigated whether the use of procalcitonin testing, to guide antibiotic prescribing, safely reduced antibiotic use amongst hospitalised patients with COVID-19 during the first wave of the pandemic using routinely collected patient institutional clinical databases and patient medical records. Data were collected in 11 National Health Service (NHS) acute hospital Trusts and Health Boards in England and Wales, and data in a pseudo-anonymised format was received from the Cardiff Clinical Trials Unit who were the data controllers for the PEACH study.

Workstream 2 will compare the oral resistome of patients with and without penicillin allergy. Metagenomic and metatranscriptomic analysis will be used for resistome assessment.

Workstream 3 will determine the feasibility of investigating if antibiotic resistance genes are lost after removal of an incorrect penicillin allergy record. This workstream will recruit patients enrolled in the Allergy Antibiotics and Microbial Resistance (ALABAMA) trial (NCT04108637), which is a randomised control trial (RCT) designed to assess the effect of removing incorrect penicillin allergy records on health outcomes. Participants are randomised to either usual care or the intervention group where they receive a novel penicillin allergy assessment pathway (PAAP), if patients in the intervention group are found to be not allergic to penicillin, their allergy label is subsequently removed. Patients recruited to this workstream will be followed up as per the ALABAMA protocol but will also be required to provide baseline and follow up (> 6 months after enrolment or allergy testing) saliva +/- stool samples. Metagenomic and metatranscriptomic analysis will be used for resistome assessment.

ELIGIBILITY:
Inclusion Criteria:

* Workstream 1

  1. Adult (>16 years) with confirmed COVID-19 (positive PCR test)
  2. Admitted to participating NHS Trusts/hospitals between 01/02/2020 to 30/06/2020
* Workstream 2

  1. Adult (≥18 years) patients with a penicillin allergy or a matched patients (by age and sex) without a penicillin allergy
  2. Received antibiotics in the 24 months prior to recruitment
  3. Willing to provide saliva +/- stool samples
* Workstream 3

  1. Patients enrolled into the ALABAMA trial

Exclusion Criteria:

* Workstream 1

  a. Patients with their allergy status missing will be excluded.
* Workstream 2

  1. Patients unable to give informed consent or who are unwilling/unable to provide saliva samples
  2. Unwilling/unable to provide saliva samples
* Workstream 3

  1. Patients unable to give informed consent or who are unwilling/unable to provide saliva samples
  2. Unwilling/unable to provide saliva samples

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: - Workstream 1 population: Participants included in the Procalcitonin Evaluation of Antibiotic use in COVID-19 Hospitalised patients (PEACH) study (ISRCTN66682918)
  - Workstream 2 population: Participants will be recruited from patients attending outpatient clinics at Leeds Teaching Hospitals NHS Trust, United Kingdom.
  - Workstream 3 population: Participants will be recruited from the population of patients participating in the he Allergy Antibiotics and Microbial Resistance (ALABAMA) trial (NCT04108637).
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Workstream 1: 60 day mortality in patients with and without penicillin allergy | 60 days from the date of positive COVID 19 test
  This outcome will measure mortality within 60 days of positive COVID-19 test. Comparative analysis will be conducted between patients with and without a documented penicillin allergy.
Workstream 2: The prevalence of antibiotic resistance genes (ARGs) in the mouth of patients with and without a penicillin allergy record. | At enrolment
  The prevalence of ARGs will be assessed using shotgun metagenomic sequencing of saliva samples. Comparative analysis will be conducted between patients with and without a documented penicillin allergy.
Workstream 3: Change in abundance of antibiotic resistance genes in saliva samples collected from participants enrolled in the ALABAMA trial | At enrolment (first sample collection) and 6 to 12 months post-enrolment (second sample collection)
  This outcome will determine the change in antibiotic resistance gene (ARG) abundance over time in patients who received the ALABAMA trial intervention (penicillin allergy assessment) compared to those in the control group (no penicillin allergy assessment). This analysis will focus on the subset of ALABAMA trial patients with at least one antibiotic prescription prior to their second saliva sampling. Comparative analysis will be conducted between the penicillin allergy assessment group and the no penicillin allergy assessment group.

SECONDARY OUTCOMES:
Workstream 1: Length of hospital stay in patients with and without a penicillin allergy. | Time of hospital admission to discharge or inpatient death for each patient, assessed up to 600 days
  This will be determined by a retrospective measurement of total hospital stay (day 0 = date of admission), calculated as days from admission date to the date of discharge or inpatient death (whichever occurred first). Comparative analysis will be conducted between patients with and without a documented penicillin allergy.
Workstream 1: Number of AMR bacterial infections in patients with and without a penicillin allergy. | Time of hospital admission to discharge or inpatient death for each patient, assessed up to 600 days
  This will be determined by blood cultures and deep respiratory culture positivity, and a infection will be considered to be a AMR/resistant infection if the isolated pathogen is resistant to ≥1 antibiotic agent in 3 or more antibiotic classes. Comparative analysis will be conducted between patients with and without a documented penicillin allergy.
Workstream 1: Total antibiotic usage in patients with and without a penicillin allergy. | Time of hospital admission to discharge or inpatient death for each patient, assessed up to 600 days
  This outcome will assess inpatient antibiotic use including antibiotic agent, route of administration and duration following COVID-19 diagnosis in hospital from day 1 of COVID-19 diagnosis to date of discharge or death (inclusive of day 1 and last day). Comparative analysis will be conducted between patients with and without a documented penicillin allergy.
Workstream 1: Rates of treatment failure in patients with and without a penicillin allergy. | Time of hospital admission to discharge or inpatient death for each patient, assessed up to 600 days
  This will be defined as re-prescription of an antibiotic within 30 days of index antibiotic prescription. Comparative analysis will be conducted between patients with and without a documented penicillin allergy.
Workstream 1: ICU admission rates in patients with and without a penicillin allergy. | Time of hospital admission to discharge or inpatient death for each patient, assessed up to 600 days
  The number of admission to intensive care units (ICU) will be counted. Comparative analysis will be conducted between patients with and without a documented penicillin allergy.
Workstream 1: Rate of Clostridioides difficile infection in patients with and without a penicillin allergy. | Time of hospital admission to discharge or inpatient death for each patient, assessed up to 600 days
  This will be determined by a toxin positive result from day 1 of COVID-19 diagnosis. Comparative analysis will be conducted between patients with and without a documented penicillin allergy.
Workstream 1: 30 day mortality in patients with and without a penicillin allergy | 30 days from COVID-19 diagnosis
  This outcome will measure mortality within 30 days of COVID-19 diagnosis in patients with and without penicillin allergy.
Workstream 2: The difference in diversity of antibiotic resistance genes (ARGs) in oral microbiome of patients with and without a penicillin allergy record. | Enrolment
  This outcome will assess the diversity of ARGs using shotgun metagenomic and metatranscriptomic sequencing of saliva samples collected at the time of enrolment. Bioinformatic analysis will be performed to quantify the overall counts, relative abundance, and diversity indices (e.g., Shannon and Simpson diversity) of ARGs. Comparative analysis will be conducted between patients with and without penicillin allergy to determine differences in ARG diversity.
Workstream 2: The number of resistance genes to specific antibiotic classes present in the oral microbiome of patients with and without a penicillin allergy record. | Enrolment
  This outcome will assess the number antibiotic resistance genes (ARGs) associated with specific antibiotic classes using shotgun metagenomic sequencing of saliva samples. A comparative analysis will be conducted between patients with and without a documented penicillin allergy.
Workstream 2: To determine whether a metagenomic or transcriptomic approach could be used to predict phenotypic antibiotic susceptibility | Enrolment
  This outcome will evaluate whether of shotgun metagenomic and metatranscriptomic sequencing of saliva samples can be used to predict phenotypic antibiotic susceptibility. Saliva samples taken at enrolment will undergo metagenomic and transcriptomic sequencing analysis to identify antibiotic resistance genes and their expression as well as antimicrobial susceptibility testing (AST) on cultured bacterial isolates from the same samples to determine actual resistance profiles.
Workstream 3: The change in the abundance and richness of antibiotic resistance genes (ARGs) over time between patients who had the ALABAMA trial intervention and those in the control group | At enrolment (first sample collection) and 6 to 12 months post-enrolment (second sample collection).
  This outcome will assess the change over time in the abundance and richness of ARGs in the oral microbiome, and where available, the gut microbiome. Samples will be analysed using shotgun metagenomic sequencing of saliva and optional stool samples. Bioinformatic analysis will include overall ARG counts, relative abundance and diversity indices (e.g., Shannon and Simpson diversity).
  Comparative analysis will be conducted between patients who received the intervention (penicillin allergy assessment) and those in the control group (no penicillin allergy assessment) to evaluate differences in ARG dynamics over time.
Workstream 3: The number and abundance of 'non-penicillin' antibiotic resistance genes in patients who had the ALABAMA trial intervention (penicillin allergy assessment) and those in the control group (no penicillin allergy assessment). | At enrolment (first sample collection) and 6 to 12 months post-enrolment (second sample collection)
  This outcome will assess the number and abundance of ARGs associated with non-penicillin antibiotic classes (e.g., macrolides, tetracyclines, fluoroquinolones, aminoglycosides) in the oral microbiome, and where available, the gut microbiome. Comparative analysis will be conducted between patients who received the intervention and those in the control group to evaluate differences in ARG dynamics over time.
Workstream 3: The number and abundance of 'penicillin' antibiotic resistance genes (ARGs) in patients who had the ALABAMA trial intervention (penicillin allergy assessment) and those in the control group (no penicillin allergy assessment). | At enrolment (first sample collection) and 6 to 12 months post-enrolment (second sample collection).
  This outcome will assess the number and abundance of ARGs specifically associated with penicillin-class antibiotics in the oral microbiome, and where available, the gut microbiome. Comparative analysis will be conducted between patients who received the intervention and those in the control group to evaluate differences in ARG dynamics over time.

OTHER OUTCOMES:
Workstream 3: To determine the number of patients from the ALABAMA trial who consented to participate in this sub-study. | From the start of recruitment until the end of the recruitment period, estimated to last up to 5 years
  Feasibility outcome to evaluate the feasibility of conducting the ARG sub-study by reporting the number and percentage of ALABAMA trial participants who provided consent to join the sub-study.
Workstream 3: To determine the number of patients who provide baseline samples | At enrolment
  Feasibility outcome to evaluate the feasibility of conducting the ARG sub-study by reporting the number and percentage of participants who provide a sample at baseline (enrolment).
Workstream 3: To determine the number of patients who provide a second sample | Six to twelve months post-enrolment
  Feasibility outcome to evaluate the feasibility of conducting the ARG sub-study by reporting the number and percentage of participants who provide a second sample 6 to 12 months post-enrolment.
Workstream 3: Explore the relationship between antibiotic resistance gene (ARG) abundance and treatment response failure | Up to 12 months post-enrolment
  This feasibility outcome aims to generate initial data to inform the design of future research studies. Measures will include relative abundance of ARGs.
Workstream 3: Explore the relationship between antibiotic resistance gene (ARG) richness and treatment response failure | Up to 12 months post-enrolment
  This feasibility outcome aims to generate initial data to inform the design of future research studies. Measures will include overall counts of unique ARGs and diversity indices to assess ARG richness.

CONTACTS AND LOCATIONS:
Overall Officials: Shadia Ahmed, MBChB, Principal Investigator — Univeristy of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS trust, Leeds, United Kingdom

DOCUMENTS (2):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT07177690/Prot_000.pdf
  • Statistical Analysis Plan (2025-07-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT07177690/SAP_001.pdf